CLINICAL TRIAL: NCT05414734
Title: A Single and Multiple Assending Doses Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamic Characteristics and Food Effect After Administration of HHT120 Capsule in Healthy Subjects
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Characteristics of HHT120 in Healthy Subjects
Acronym: HHT120
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Commercialization consideration. Without safety issues.
Sponsor: Shanghai Synergy Pharmaceutical Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DTYX21037PⅠ
Record Dates: First submitted 2022-05-27; First posted 2022-06-10 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SAD HHT120 (Experimental): Subjects will receive a single dose of HHT120 from 7 doses.
  Interventions: Drug: HHT120
- SAD Placebo (Placebo Comparator): Subjects will receive a single dose of matched Placebo.
  Interventions: Drug: Placebo
- MAD HHT120 (Experimental): Subjects will receive a mutiple-dose of HHT120 twice daily for 7 days from 3 doses.
  Interventions: Drug: HHT120
- MAD Placebo (Placebo Comparator): Subjects will receive a mutiple-dose of matched placebo twice daily for 7 days.
  Interventions: Drug: Placebo
- FE K-C (Experimental): Subjects will receive a single dose of HHT120 in the morning in fasted condition in Period 1; followed by a single dose of HHT120 administered in the morning in fed condition in Period 2. A washout period of 7 days will be maintained between 2 periods.
  Interventions: Drug: HHT120
- FE C-K (Experimental): Subjects will receive a single dose of HHT120 in the morning in fed condition in Period 1; followed by a single dose of HHT120 administered in the morning in fasted condition in Period 2. A washout period of 7 days will be maintained between 2 periods.
  Interventions: Drug: HHT120

INTERVENTIONS:
Drug: HHT120 — Capsule, oral administration
  Other Names: PTI-011-Cl
  Arms: FE C-K; FE K-C; MAD HHT120; SAD HHT120
Drug: Placebo — Capsule, oral administration
  Arms: MAD Placebo; SAD Placebo

SUMMARY:
This is a first in human clinical trial with HHT120. The purpose of this study is to characterize the safety, pharmacokinetic (PK) and Pharmacodynamic (PD) profile of single and multiple twice-daily doses of HHT120 in healthy Subjects and to assess the effects of food on the PK profile of single-dose of HHT120 in healthy Subjects.

DETAILED DESCRIPTION:
There are 3 parts of the study:

Part 1: Single asending dose trial; Part 2: Multiple asending dose trial; Part 3: Food effect trial ( 2-Period Crossover)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and are willing to follow the clinical trial protocol to complete the study and sign the informed consent voluntarily
2. ≥50 kg, BMI 19.0-26.0 kg/m2 (including the critical value);
3. Those who have been proved healthy by medical history inquiry, physical examination and laboratory examination.

Exclusion Criteria:

1. Have a blood coagulation dysfunction or bleeding tendency, such as repeated bleeding gums, or nearly six months increased risk of bleeding events, or platelet count < 100 x 109 / L, or always have intracranial hemorrhage (after the accident, for example), gastrointestinal bleeding, purpura, or with active pathological bleeding, bleeding or have any family history, etc.
2. History of motor system, nervous/psychiatric system, endocrine system, blood circulation system, respiratory system, digestive system, urinary system, reproductive system abnormalities or existing diseases mentioned above, which the researcher judged to be clinically significant;
3. History of drug or food allergy, or are allergic to the active ingredients of the test drug and any excipient ingredients;
4. History of postural hypotension, fainting or coma;
5. High risk factors of TdP (hypokalemia, hypomagniemia, bradycardia, heart failure, hereditary long QT syndrome, etc.);
6. QTc interval greater than 450ms during screening;
7. Undergone surgery within 3 months prior to or during screening, or have undergone surgery that affects drug absorption, distribution, metabolism or excretion, or plan to undergo surgery during the study period;
8. Blood donation or massive blood loss (≥400 mL) within 3 months before screening or during screening (except female menstrual period);
9. History of drug abuse or positive urine drug screening (morphine, THC, methylamphetamine, dimethylene dioxy-amphetamine, ketamine) within 5 years before screening;
10. Excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups per day, 1 cup =250 mL) within 3 months prior to screening or during screening;
11. Drank regularly within 3 months prior to screening or during screening, i.e. drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45mL 40% alcohol spirits or 150mL wine), who could not abstain from drinking during the test, or whose alcohol breath test results were > 0 mg/100mL;
12. Smoking ≥5 cigarettes per day in the previous 3 months in the screening period; Or unable to stop using any tobacco products in the treatment period;
13. Consumed a large amount of drinks or food (such as grapefruit, grapefruit juice, grapefruit jam, etc.) rich in grapefruit, pomelo, star fruit, mango and dragon fruit within the previous 14 days prior to screening; Or any beverage or food containing grapefruit (i.e. grapefruit), pomelo, star fruit, mango, dragon fruit within 48 hours before the first dose;
14. Special dietary requirements, unable to follow the uniform diet or dysphagia;
15. Lactose intolerant (who had diarrhea after drinking milk);
16. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health care products within 14 days prior to screening;
17. Received vaccination within 28 days prior to or during screening;
18. Have participated in other clinical trials within 3 months prior to or during screening or who are not themselves participating in clinical trials;
19. Pregnant or lactating women, or abnormal pregnancy tests that are clinically significant as determined by the investigator; Male subjects (or their partners) or female subjects who have planned to have children during the entire study period and within 6 months after the study end and are unwilling to use one or more non-drug contraceptive methods (e.g., complete abstinence, condoms, vasectomy, etc.) during the study period;
20. Female subjects with irregular menstruation or menstrual disorder (including menstrual cycle disorder, menstrual disorder and menorrhagia);
21. Those who cannot tolerate venipuncture or have difficulty in collecting blood;
22. Abnormal physical examination, blood routine examination, blood biochemistry, coagulation function, urine routine examination, 12-lead electrocardiogram examination, chest X-ray examination and clinical significance determined by the investigator;
23. Abnormal vital signs and abnormal retest;
24. Hepatitis B surface antigen, treponema pallidum antibody, human immunodeficiency virus antibody and hepatitis C antibody are abnormal and clinically significant as determined by researchers;
25. The investigator considers that the subjects are not suitable to participate in the study for other reasons or the subjects withdraw from the study for their own reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Vital signs | Up to Day 14
  Abnormal changes in vital signs from baseline
Physical examination | Up to Day 14
  Abnormal changes in physical examination from baseline
Laboratory examination | Up to Day 14
  Abnormal changes in laboratory examination from baseline
Electrocardiogram | Up to Day 14
  Abnormal changes in electrocardiogram from baseline
Chest radiography | Up to Day 14
  Abnormal changes in chest radiography from baseline
Adverse events | Up to Day 14
  Incidence of adverse events, serious adverse events, adverse events of special interest
Maximum tolerable dose (MTD) | Up to Day 14
  Maximum tolerable dose (MTD)

SECONDARY OUTCOMES:
Part 1: Cmax | Up to Day 4
  Cmax of single dose administration
Part 1: Tmax | Up to Day 4
  Tmax of single dose administration
Part 1: t1/2 | Up to Day 4
  t1/2 of single dose administration
Part 1: Vz/F | Up to Day 4
  Vz/F of single dose administration
Part 1: CLz/F | Up to Day 4
  CLz/F of single dose administration
Part 1: AUC | Up to Day 4
  AUC of single dose administration
Part 2: Cmax,ss | Up to Day 10
  Cmax,ss of multiple dose administration
Part 2: AUC,ss | Up to Day 10
  AUC,ss of multiple dose administration
Part 2: Tmax,ss | Up to Day 10
  tmax,ss of multiple dose administration
Part 2: Cmin,ss | Up to Day 10
  Cmin,ss of multiple dose administration
Part 2: Cav,ss | Up to Day 10
  Cav,ss of multiple dose administration
Part 2: t1/2 | Up to Day 10
  t1/2 of multiple dose administration
Part 2: MRTss | Up to Day 10
  MRTss of multiple dose administration
Part 2: Accumulation index | Up to Day 10
  accumulation index of multiple dose administration
Part 1 & Part 2: aPTT, INR and TT | Up to Day 10
  Maximum percentage of aPTT, INR and TT to baseline (Emax)
Part 3: Cmax in fasted or fed condition | Up to Day 4
  Geometric mean ratios of Cmax (fed/fasted) and their 90% confidence intervals
Part 3: AUC in fasted or fed condition | Up to Day 4
  Geometric mean ratios of AUC (fed/fasted) and their 90% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Yiqing Zhao, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China